CLINICAL TRIAL: NCT00193362
Title: Phase III Randomized Study of Paclitaxel, Carboplatin, and Gemcitabine Versus Gemcitabine and Vinorelbine as First-Line Chemotherapy for Stage IIIB and IV Non-Small Cell Lung Cancer
Brief Title: Study of Paclitaxel, Carboplatin, and Gemcitabine Versus Gemcitabine and Vinorelbine for Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Eli Lilly and Company (Industry); GlaxoSmithKline (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI LUN 54; B9E-MC-X338; VNR-R47
Record Dates: First submitted 2005-09-12; First posted 2005-09-19 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Paclitaxel; Carboplatin; Gemcitabine; Vinorelbine

INTERVENTIONS:
Drug: Paclitaxel
Drug: Carboplatin
Drug: Gemcitabine
Drug: Vinorelbine

SUMMARY:
The purpose of this study is to compare the effectiveness of the three-drug combination paclitaxel, carboplatin, and gemcitabine to the two-drug combination gemcitabine and vinorelbine in patients with advanced Non-Small Cell Lung Cancer

DETAILED DESCRIPTION:
Upon determination of eligibility, patients will be randomly assigned to one of two treatment arms:

* Paclitaxel + Carboplatin + Gemcitabine
* Gemcitabine + Vinorelbine

For ever 2 patients treated, 1 will receive treatment A (Paclitaxel + Carboplatin + Gemcitabine) and 1 will receive treatment B (Gemcitabine + Vinorelbine). The study is not blinded so both the patient and the doctor will know which treatment has been assigned.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, you must meet the following criteria:

* Non-small cell bronchogenic carcinoma
* Newly diagnosed unresectable stage IIIB or stage IV disease
* Patients with stage IIIB disease should be ineligible for combined therapy
* Patients must have measurable lesion definable by X-ray or CT scan.
* No prior antineoplastic chemotherapy for lung cancer prior to study entry
* Age > 18 years
* Able to perform activities of daily living with minimal assistance
* Adequate bone marrow, liver and kidney function
* Written informed consent must be obtained prior to study entry
* Patients must be available for treatment and followup.

Exclusion Criteria:

You cannot participate in this study if any of the following apply to you:

* Female patient pregnant or lactating
* History of heart disease
* Serious active infection at the time of treatment
* Other serious underlying medical condition
* Brain metastasis
* Patients without measurable disease
* Uncontrolled diabetes mellitus defined as random blood sugar > 250mg/dL
* Dementia or significantly altered mental status
* Significant peripheral neuropathy by history or physical examination.

Please note: There are additional inclusion/exclusion criteria. The study center will determine if you meet all of the criteria. If you do not qualify for the trial, study personnel will explain the reasons. If you do qualify, study personnel will explain the trial in detail and answer any questions you may have.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200
Dates: Start 2004-06; Primary Completion 2005-06 (Actual); Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Overall survival.

SECONDARY OUTCOMES:
Overall toxicity
Overall response rate
Time-to-progression
Assess the quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Greco, MD, Principal Investigator — SCRI Development Innovations, LLC

REFERENCES:
- [Result] Greco FA, Spigel DR, Kuzur ME, Shipley D, Gray JR, Thompson DS, Burris HA, Yardley DA, Pati A, Webb CD, Gandhi JG, Hainsworth JD. Paclitaxel/Carboplatin/gemcitabine versus gemcitabine/vinorelbine in advanced non-small-cell lung cancer: a phase II/III study of the Minnie Pearl Cancer Research Network. Clin Lung Cancer. 2007 Sep;8(8):483-7. doi: 10.3816/CLC.2007.n.032. PMID 17922972
- See also: Published article in Clinical Lung Cancer — http://cigjournals.metapress.com/content/j662866rh7152581/?p=38ed22b862d2470fb98c82b3d3c7dc94&pi=3